CLINICAL TRIAL: NCT01389323
Title: Open-Label, Single Arm Evaluation of BMS-790052 (Daclatasvir) in Combination With Peg-Interferon Alfa-2a and Ribavirin in Black-African Americans, Latinos and White-Caucasians With Chronic Hepatitis C Genotype 1 Infection
Brief Title: BMS-790052 (Daclatasvir) Plus Peg-Interferon Alfa-2a and Ribavirin in Treatment-Naive Black/African-Americans, Latinos and White/Caucasians With Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI444-038
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: Daclatasvir + Peg-Interferon Alfa-2a + Ribavirin (Experimental)
  Interventions: Drug: Daclatasvir; Drug: Peg-Interferon Alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Daclatasvir — Tablet, Oral, 60 mg, once daily, 24 weeks
  Other Names: BMS-790052
Drug: Peg-Interferon Alfa-2a — Syringe, Subcutaneous Injection, 180 μg, Once weekly, 24 or 48 weeks depending on response
  Other Names: Pegasys
Drug: Ribavirin — Tablet, Oral, 1000 or 1200 mg based on weight, Twice daily, 24 or 48 weeks depending on response
  Other Names: Copegus

SUMMARY:
The purpose of this study is to compare the rates of sustained virologic response in each cohort (Black-African Americans, Latinos) in this study to historical rate.

ELIGIBILITY:
Inclusion Criteria:

* Participants chronically infected with Hepatitis C virus (HCV) genotype 1
* HCV RNA viral load of ≥10,000 IU/mL at screening
* No previous exposure to interferon formulation, ribavirin or HCV direct antiviral agent
* Self-described as Black-African American, Latino or White-Caucasian
* Results of a liver biopsy obtained ≤36 months prior to first treatment compensated cirrhotics with HCV liver biopsy from any time prior to first treatment.

Compensated cirrhotics were capped at approximately 25%

Exclusion Criteria:

* Evidence of decompensated liver disease
* Documented or suspected Hepatocellular carcinoma (HCC)
* Positive for Hepatitis B or HIV 1/HIV 2 antibody at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (36):
- United States (35):
  - Alabama Liver & Digestive Specialists (Alds), Montgomery, Alabama
  - Va Long Beach Healthcare System - 11, Long Beach, California
  - Axis Clinical Trials, Los Angeles, California
  - Greater Los Angeles Healthcare System, Los Angeles, California
  - University Of California, Davis Medical Center, Sacramento, California
  - Ucsd Antiviral Research Center (Avrc), San Diego, California
  - Precision Research Institute, Llc, San Diego, California
  - Medical Associates Research Group, Inc, San Diego, California
  - Miami V.A. Healthcare System, Maimi, Florida
  - University Of Miami, Miami, Florida
  - Florida Hospital Transplant Center, Orlando, Florida
  - Infectious Disease Research Institute, Inc, Tampa, Florida
  - South Florida Center Of Gastroenterology, P.A., Wellington, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Atlanta Medical Center, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Digestive Disease Associates, P.A., Baltimore, Maryland
  - The Research Institute, Springfield, Massachusetts
  - Digestive Health Center, Ocean Springs, Mississippi
  - Montefiore Medical Center, The Bronx, New York
  - University Of North Carolina At Chapel Hill School Of Med, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Carolinas Center For Liver Disease, Statesville, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Texas Clinical Research Institute, Arlington, Texas
  - Baylor College Of Medicine, Houston, Texas
  - Liver Associates Of Texas, Houston, Texas
  - Research Specialists Of Texas, Houston, Texas
  - Texas Liver Institute, San Antonio, Texas
  - Brooke Army Medical Center, San Antonio, Texas
  - Metropolitan Research, Annandale, Virginia
  - Mcguire D V A M C, Richmond, Virginia
- Local Institution, San Juan, Puerto Rico

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 33 clinical sites in United States.
Pre-assignment Details: A total of 448 participants were enrolled, and 246 entered treatment period. Remaining 202 did not enter treatment period (29: withdrew consent, 17: lost to follow-up, 156: no longer met study criteria). As per protocol, any participant who discontinued the treatment period was still expected to enter the post-treatment follow-up period.
Groups:
- Daclatasvir + Pegylated-interferon Alfa 2a + Ribavirin: Participants received daclatasvir (BMS-790052) 60 mg tablet orally once daily, along with pegylated-interferon alfa 2a solution for injection 180 μg/0.5 mL subcutaneously once weekly, and ribavirin 1000 mg per day for those weighing <75 kg or 1200 mg per day for those weighing ≥75 kg for a period of 24 weeks. Participants who achieved a virologic response (Hepatitis C Virus RNA undetectable at both Weeks 4 and 12) completed therapy at Week 24 and were followed for 48 weeks of post-treatment follow-up. Participants who did not achieve the virologic response, continued to receive pegylated-interferon alfa 2a and ribavirin for additional 24 weeks (total treatment duration of 48 weeks), and were followed for 24 weeks of post-treatment follow-up. Dose modifications to pegylated-interferon alfa 2a and ribavirin were allowed to manage tolerability and adverse events.
Period: Treatment Period (up to 48 Weeks)
Arm/Group | Daclatasvir + Pegylated-interferon Alfa 2a + Ribavirin
Started | 246
Completed | 151
Not Completed | 95
Not completed — Lack of Efficacy | 41
Not completed — Adverse Event | 24
Not completed — Participant's request to discontinue | 6
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 10
Not completed — Poor/non-compliance | 5
Not completed — Did not meet study criteria | 2
Period: Follow-up Period (up to 48 Weeks)
Arm/Group | Daclatasvir + Pegylated-interferon Alfa 2a + Ribavirin
Started | 221 (Out of 246 participants who entered the treatment period, 221 continued in the follow-up period.)
Completed | 184
Not Completed | 37
Not completed — Withdrawal by Subject | 10
Not completed — Lost to Follow-up | 22
Not completed — Follow-up no longer needed per protocol | 2
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Population: All treated participants.
Arm/Group | Daclatasvir + Pegylated-interferon Alfa 2a + Ribavirin
Number analyzed (Participants) | 246
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 177
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 107
  Not Hispanic or Latino | 139
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 128
  White | 118
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black/African American Latino | 19
  Black/African American Non-Latino | 109
  White Latino | 88
  White/Caucasian Non-Latino | 30
Hepatitis C Virus RNA Levels [Mean (Standard Deviation); unit: Log10 IU/mL] | 6.21 (0.684)
Hepatitis C Virus RNA Distribution [Number; unit: participants]
  <800,000 IU/mL | 64
  ≥800,000 IU/mL | 182
Hepatitis C Virus Genotype [Number; unit: participants]
  Subtype 1A | 191
  Subtype 1B | 54
  Subtype 1 | 1
rs12979860 Single Nucleotide Polymorphism in the Interleukin-28B Gene [Number; unit: participants]
  Wild Type (CC) | 50
  Heterozygous (CT) | 134
  Minor Homozygous (TT) | 62

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response at Post-treatment Week 12 (SVR12)
Description: SVR12 was defined as Hepatitis C Virus (HCV) RNA levels <lower limit of quantitation (LLOQ), (target detected or target not detected) at Post-treatment Week 12. The limit of detection for HCV RNA was 10 IU/mL and the LLOQ was 25 IU/mL. For analysis purpose, participants were assigned to following 3 race/ethnicity cohorts: Black/African American, Latino, and White non-Latino. Some participants were represented in more than one race/ethnicity cohort.
Time Frame: Post-treatment Week 12
Population: All treated participants. Modified intent-to-treat analysis (participants meeting the response criteria / all treated participants) was performed for Black/African American and Latino cohorts.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Black/African American Cohort: Participants belonging to Black/African American race, received daclatasvir (BMS-790052) 60 mg tablet orally once daily, along with pegylated-interferon alfa 2a solution for injection 180 μg/0.5 mL subcutaneously once weekly, and ribavirin 1000 mg per day for those weighing <75 kg or 1200 mg per day for those weighing ≥75 kg for a period of 24 weeks. Participants who achieved a virologic response (HCV RNA undetectable at both Weeks 4 and 12) completed therapy at Week 24 and were followed for 48 weeks of post-treatment follow-up. Participants who did not achieve the virologic response, continued to receive pegylated-interferon alfa 2a and ribavirin for additional 24 weeks (total treatment duration of 48 weeks), and were followed for 24 weeks of post-treatment follow-up. Dose modifications to pegylated-interferon alfa 2a and ribavirin were allowed to manage tolerability and adverse events (AEs). This cohort included Latino and Non-Latino participants.
- Latino Cohort: Participants belonging to Latino ethnicity, received daclatasvir (BMS-790052) 60 mg tablet orally once daily, along with pegylated-interferon alfa 2a solution for injection 180 μg/0.5 mL subcutaneously once weekly, and ribavirin 1000 mg per day for those weighing <75 kg or 1200 mg per day for those weighing ≥75 kg for a period of 24 weeks. Participants who achieved a virologic response (HCV RNA undetectable at both Weeks 4 and 12) completed therapy at Week 24 and were followed for 48 weeks of post-treatment follow-up. Participants who did not achieve the virologic response, continued to receive pegylated-interferon alfa 2a and ribavirin for additional 24 weeks (total treatment duration of 48 weeks), and were followed for 24 weeks of post-treatment follow-up. Dose modifications to pegylated-interferon alfa 2a and ribavirin were allowed to manage tolerability and AEs. This cohort included White/Caucasian and Black/African American participants.
- White Non-Latino Cohort: Participants belonging to White race and Non-Latino ethnicity, received daclatasvir (BMS-790052) 60 mg tablet orally once daily, along with pegylated-interferon alfa 2a solution for injection 180 μg/0.5 mL subcutaneously once weekly, and ribavirin 1000 mg per day for those weighing <75 kg or 1200 mg per day for those weighing ≥75 kg for a period of 24 weeks. Participants who achieved a virologic response (HCV RNA undetectable at both Weeks 4 and 12) completed therapy at Week 24 and were followed for 48 weeks of post-treatment follow-up. Participants who did not achieve the virologic response, continued to receive pegylated-interferon alfa 2a and ribavirin for additional 24 weeks (total treatment duration of 48 weeks), and were followed for 24 weeks of post-treatment follow-up. Dose modifications to pegylated-interferon alfa 2a and ribavirin were allowed to manage tolerability and AEs.
Arm/Group | Black/African American Cohort | Latino Cohort | White Non-Latino Cohort
Number analyzed (Participants) | 128 | 107 | 30
percentage of participants | 50.8 [42.1 to 59.4] | 57.0 [47.6 to 66.4] | 66.7 [49.8 to 83.5]

2. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response at Post-treatment Week 12 (SVR12) With rs12979860 Single Nucleotide Polymorphisms at Baseline in the Interleukin-28B Gene
Description: as for outcome 1
Time Frame: Post-treatment Week 12
Population: All treated participants. Here, 'n' signifies the number of participants evaluable in the specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Black/African American Cohort | Latino Cohort | White Non-Latino Cohort
Number analyzed (Participants) | 128 | 107 | 30
percentage of participants
  Wild Type (CC) (n=20, 24, 10) | 80.0 [62.5 to 97.5] | 70.8 [52.6 to 89.0] | 80.0 [55.2 to 100.0]
  Heterozygous (CT) (n=58, 69, 17) | 53.4 [40.6 to 66.3] | 50.7 [38.9 to 62.5] | 58.8 [35.4 to 82.2]
  Minor Homozygous (TT) (n=50, 14, 3) | 36.0 [22.7 to 49.3] | 64.3 [39.2 to 89.4] | 66.7 [13.3 to 100.0]

3. Secondary Outcome: Percentage of Participants With Hepatitis C Virus (HCV) RNA Levels <Lower Limit of Quantitation (LLOQ), Target Detected or Target Not Detected, at Specified Time Points
Description: The limit of detection for HCV RNA levels was 10 IU/mL and the LLOQ was 25 IU/mL. Data for post-treatment Weeks 36 and 48 were based on participants who had achieved virologic response (defined as HCV RNA levels <LLOQ, target not detected) at both Weeks 4 and 12, and completed 24 weeks of study treatment. For analysis purpose, participants were assigned to following 3 race/ethnicity cohorts: Black/African American, Latino, and White non-Latino. Some participants were represented in more than one race/ethnicity cohort.
Time Frame: Weeks 1, 2, 4, 6, 8, 12; both Weeks 4 and 12; end-of-treatment (up to 48 weeks), or post-treatment Week 24
Population: All treated participants. Here, 'N' (number of participants analyzed) signifies number of participants evaluable at the specified time-points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Black/African American Cohort | Latino Cohort | White Non-Latino Cohort
Number analyzed (Participants) | 128 | 107 | 30
percentage of participants
  Week 1 | 32.8 [24.7 to 40.9] | 44.9 [35.4 to 54.3] | 33.3 [16.5 to 50.2]
  Week 2 | 64.1 [55.8 to 72.4] | 72.0 [63.5 to 80.5] | 60.0 [42.5 to 77.5]
  Week 4 | 77.3 [70.1 to 84.6] | 85.0 [78.3 to 91.8] | 66.7 [49.8 to 83.5]
  Week 6 | 76.6 [69.2 to 83.9] | 81.3 [73.9 to 88.7] | 80.0 [65.7 to 94.3]
  Week 8 | 76.6 [69.2 to 83.9] | 81.3 [73.9 to 88.7] | 76.7 [61.5 to 91.8]
  Week 12 | 71.1 [63.2 to 78.9] | 80.4 [72.8 to 87.9] | 76.7 [61.5 to 91.8]
  Both Weeks 4 and 12 | 68.0 [59.9 to 76.1] | 77.6 [69.7 to 85.5] | 56.7 [38.9 to 74.4]
  EOT | 73.4 [65.8 to 81.1] | 79.4 [71.8 to 87.1] | 93.3 [84.4 to 100.0]
  Post-treatment Week 24 | 46.9 [38.2 to 55.5] | 57.0 [47.6 to 66.4] | 63.3 [46.1 to 80.6]

4. Secondary Outcome: Percentage of Participants With Hepatitis C Virus (HCV) RNA Levels <Lower Limit of Quantitation (LLOQ), Target Not Detected, at Specified Time Points
Description: The limit of detection for HCV RNA levels was 10 IU/mL and the LLOQ was 25 IU/mL. For analysis purpose, participants were assigned to following 3 race/ethnicity cohorts: Black/African American, Latino, and White non-Latino. Some participants were represented in more than one race/ethnicity cohort.
Time Frame: Weeks 1, 2, 4, 6, 8, 12; both Weeks 4 and 12; end-of-treatment (up to 48 weeks), or post-treatment Weeks 12 and 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Black/African American Cohort | Latino Cohort | White Non-Latino Cohort
Number analyzed (Participants) | 128 | 107 | 30
percentage of participants
  Week 1 | 6.3 [2.1 to 10.4] | 12.1 [6.0 to 18.3] | 6.7 [0.0 to 15.6]
  Week 2 | 28.1 [20.3 to 35.9] | 27.1 [18.7 to 35.5] | 30.0 [13.6 to 46.4]
  Week 4 | 64.1 [55.8 to 72.4] | 68.2 [59.4 to 77.0] | 50.0 [32.1 to 67.9]
  Week 6 | 68.8 [60.7 to 76.8] | 75.7 [67.6 to 83.8] | 66.7 [49.8 to 83.5]
  Week 8 | 70.3 [62.4 to 78.2] | 73.8 [65.5 to 82.2] | 66.7 [49.8 to 83.5]
  Week 12 | 64.1 [55.8 to 72.4] | 74.8 [66.5 to 83.0] | 66.7 [49.8 to 83.5]
  Both Weeks 4 and 12 | 55.5 [46.9 to 64.1] | 58.9 [49.6 to 68.2] | 43.3 [25.6 to 61.1]
  EOT | 71.1 [63.2 to 78.9] | 78.5 [70.7 to 86.3] | 93.3 [84.4 to 100.0]
  Post-treatment Week 12 | 50.8 [42.1 to 59.4] | 55.1 [45.7 to 64.6] | 63.3 [46.1 to 80.6]
  Post-treatment Week 24 | 46.9 [38.2 to 55.5] | 55.1 [45.7 to 64.6] | 63.3 [46.1 to 80.6]

5. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Discontinuations Due to Adverse Events (AEs), Treatment-related AEs, and Who Died
Description: An AE was defined as any new unfavorable symptom, sign, or disease or worsening of a pre-existing condition that does not necessarily have a causal relationship with treatment. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity; was life-threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalization. Treatment-related AE was defined as an AE that had certain, probable, possible, or unknown relationship to study drug. For analysis purpose, participants were assigned to following 4 race/ethnicity cohorts: Black/African American, White/Caucasian, Latino and Non-Latino. Some participants were represented in more than one race/ethnicity cohort.
Time Frame: From first dose to last dose plus 7 days (treatment period [TP]) through 48 weeks after the end of TP (follow-up period [FUP])
Population: All treated participants for TP and all follow-up participants for FUP. Here, "n" signifies the number of participants evaluable in their respective study periods.
Measure: Number; unit: participants
Groups:
- Black/African American Cohort: Participants belonging to Black/African American race, received daclatasvir (BMS-790052) 60 mg tablet orally once daily, along with pegylated-interferon alfa 2a solution for injection 180 μg/0.5 mL subcutaneously once weekly, and ribavirin 1000 mg per day for those weighing <75 kg or 1200 mg per day for those weighing ≥75 kg for a period of 24 weeks. Participants who achieved a virologic response (HCV RNA undetectable at both Weeks 4 and 12) completed therapy at Week 24 and were followed for 48 weeks of post-treatment follow-up. Participants who did not achieve the virologic response, continued to receive pegylated-interferon alfa 2a and ribavirin for additional 24 weeks (total treatment duration of 48 weeks), and were followed for 24 weeks of post-treatment follow-up. Dose modifications to pegylated-interferon alfa 2a and ribavirin were allowed to manage tolerability and AEs. This cohort included Latino and Non-Latino participants.
- White/Caucasian Cohort: Participants belonging to White/Caucasian race, received daclatasvir (BMS-790052) tablets 60 mg orally, once daily, along with pegylated-interferon alfa 2a solution for injection 180 μg per 0.5 mL subcutaneously, once weekly, and ribavirin tablets 800 mg orally, twice daily, for 24 weeks (for participants who had achieved the virologic response at Weeks 4 and 12) to 48 weeks (for participants who did not achieve the virologic response at Weeks 4 and 12). For participants weighing <75 kg, the total dose of ribavirin was 1000 mg per day and for those weighing ≥75 kg, the dose was 1200 mg per day. Dose modifications to pegylated-interferon alfa 2a and ribavirin were allowed to manage tolerability and AEs. This cohort included Latino and Non-Latino participants.
- Non-Latino Cohort: Participants belonging to Non-Latino ethnicity, received daclatasvir (BMS-790052) tablets 60 mg orally, once daily, along with pegylated-interferon alfa 2a solution for injection 180 μg per 0.5 mL subcutaneously, once weekly, and ribavirin tablets 800 mg orally, twice daily, for 24 weeks (for participants who had achieved the virologic response at Weeks 4 and 12) to 48 weeks (for participants who did not achieve the virologic response at Weeks 4 and 12). For participants weighing <75 kg, the total dose of ribavirin was 1000 mg per day and for those weighing ≥75 kg, the dose was 1200 mg per day. Dose modifications to pegylated-interferon alfa 2a and ribavirin were allowed to manage tolerability and AEs. This cohort included White/Caucasian and Black/African American participants.
- Overall Population: Participants received daclatasvir (BMS-790052) tablets 60 mg orally, once daily, along with pegylated-interferon alfa 2a solution for injection 180 μg per 0.5 mL subcutaneously, once weekly, and ribavirin tablets 800 mg orally, twice daily, for 24 weeks (for participants who had achieved the virologic response at Weeks 4 and 12) to 48 weeks (for participants who did not achieve the virologic response at Weeks 4 and 12). For participants weighing <75 kg, the total dose of ribavirin was 1000 mg per day and for those weighing ≥75 kg, the dose was 1200 mg per day. Dose modifications to pegylated-interferon alfa 2a and ribavirin were allowed to manage tolerability and AEs.
Arm/Group | Black/African American Cohort | White/Caucasian Cohort | Latino Cohort | Non-Latino Cohort | Overall Population
Number analyzed (Participants) | 128 | 118 | 107 | 139 | 246
participants
  SAEs: TP (n=128,118,107,139,246) | 12 | 9 | 5 | 16 | 21
  Discontinued due to AE: TP (n=128,118,107,139,246) | 9 | 15 | 6 | 18 | 24
  Treatment-related AEs: TP (n=128,118,107,139,246) | 111 | 108 | 93 | 126 | 219
  Deaths: TP (n=128,118,107,139,246) | 0 | 0 | 0 | 0 | 0
  SAEs: FUP (n=117,104,96,125,221) | 3 | 0 | 1 | 2 | 3
  Deaths: FUP (n=117,104,96,125,221) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose to 7 days post last dose of study treatment
Description: On-treatment Period
Arm/Group | Daclatasvir + Pegylated-interferon Alfa 2a + Ribavirin
Serious Adverse Events (participants affected / at risk) | 21/246
Other Adverse Events (participants affected / at risk) | 227/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir + Pegylated-interferon Alfa 2a + Ribavirin (N=246)
Colitis (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 5
Drug abuse (Psychiatric disorders) | 1
Gangrene (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Osteomyelitis (Infections and infestations) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Substance abuse (Psychiatric disorders) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Syncope (Nervous system disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Gastroenteritis (Infections and infestations) | 1
Paraesthesia (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Cellulitis (Infections and infestations) | 1
Overdose (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir + Pegylated-interferon Alfa 2a + Ribavirin (N=246)
Anxiety (Psychiatric disorders) | 13
Dizziness (Nervous system disorders) | 25
Dry skin (Skin and subcutaneous tissue disorders) | 31
Influenza like illness (General disorders) | 47
Insomnia (Psychiatric disorders) | 46
Pruritus (Skin and subcutaneous tissue disorders) | 43
Back pain (Musculoskeletal and connective tissue disorders) | 16
Decreased appetite (Metabolism and nutrition disorders) | 34
Depression (Psychiatric disorders) | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23
Injection site reaction (General disorders) | 13
Neutropenia (Blood and lymphatic system disorders) | 57
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Weight decreased (Investigations) | 15
Chills (General disorders) | 35
Fatigue (General disorders) | 107
Headache (Nervous system disorders) | 77
Pain (General disorders) | 21
Vomiting (Gastrointestinal disorders) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Nausea (Gastrointestinal disorders) | 61
Anaemia (Blood and lymphatic system disorders) | 73
Diarrhoea (Gastrointestinal disorders) | 30
Irritability (Psychiatric disorders) | 26
Myalgia (Musculoskeletal and connective tissue disorders) | 18
Alopecia (Skin and subcutaneous tissue disorders) | 28
Arthralgia (Musculoskeletal and connective tissue disorders) | 24
Pyrexia (General disorders) | 23
Rash (Skin and subcutaneous tissue disorders) | 58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.